CLINICAL TRIAL: NCT02845505
Title: Intravascular Ultrasound Prediction of Myocardial Size and Coronary Computed Tomography-Derived Ischemic Burden for Coronary Lesion
Acronym: IVUS-CAMS
Status: Active, not recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Young-Hak Kim, MD, PhD, Professor, Asan Medical Center
Other Study IDs: AMCCV 2016-06
Record Dates: First submitted 2016-07-13; First posted 2016-07-27 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
Keywords: intravascular ultrasonography; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVUS-CAMS: patients who undergo coronary computed tomography angiography, invasive coronary angiography and IVUS
  Interventions: Other: Intravascular Ultrasound, coronary computed tomography angiography

INTERVENTIONS:
Other: Intravascular Ultrasound, coronary computed tomography angiography

SUMMARY:
The aims of this study are 1) to identify IVUS determinants of the CAMS-derived myocardial territories subtended to the diseased vessels, 2) to find IVUS determinant for the extent of CAMS-derived myocardial size, and 3) to develop the mathematical model that integrates the IVUS information about myocardial territory and stenosis severity and predicts the extent of CAMS-derived myocardial size.

ELIGIBILITY:
Inclusion Criteria:

* Age 20years or older
* Patients who have at least one epicardial coronary artery lesion (including isolated left main disease or side branch) with visually estimated diameter stenosis >50% and take coronary angiography, CT angiography and IVUS
* Willing and able to provide informed written consent

Exclusion Criteria:

* In-stent restenosis
* Bypass graft
* Suspected coronary spasm even after sufficient nitrate injected
* Cases in which the IVUS imaging catheter failed to cross the lesion
* Poor quality IVUS or CT images
* Visible collateral flow on angiography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergo coronary computed tomography angiography, invasive coronary angiography and IVUS assessment prior to intervention will be enrolled. The patients should have at least one coronary artery lesion (including non-left main and isolated left main disease) with visually estimated diameter stenosis >50%
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
mathematically-predicted ischemic size (by using IVUS parameters) vs. CAMS-derived myocardial size subtended to the stenotic segment | 1 year

SECONDARY OUTCOMES:
Impact of plaque characteristics (attenuated plaque, plaque rupture, calcification, thrombosis, etc.) assessed by IVUS on the ischemic burden assessed by CAMS | 1 year
Incidence of MACE comprising death, nonfatal myocardial infarction or target vessel revascularization | 1 year

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Asan Medical Center, Seoul, Songpa-Gu
  - Hallym University Sacred Heart hospital, Anyang
  - Chungnam National University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Inje university Pusan Paik hospital, Pusan
  - Kosin University Gospel Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Kangbuk Samsung Hospital, Seoul
  - Veterans Hospital Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No